CLINICAL TRIAL: NCT05282641
Title: Effects of 10-gram Collagen Protein Hydrolysate on Cardiometabolic Health in Obese (BMI 25-35 kg/m2) Men and Women With Elevated Risk to Develop Type-2 Diabetes and CVD
Brief Title: Effects of 10-gram Collagen Protein Hydrolysate on Cardiometabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: METC20-007
Record Dates: First submitted 2021-11-17; First posted 2022-03-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Glucose Metabolism; Lipid Metabolism
Keywords: Collagen hydrolysate; Glucose metabolism; Dietary patterns; Cardiometabolic health

STUDY DESIGN:
Intervention Model Description: A 4-weeks randomized, controlled trial with a parallel design. Before the 4-weeks intervention, there is a 2-weeks run period.
Who Masked: Participant, Investigator
Masking Description: The subjects will follow one of the two experimental conditions. The decision in which condition they will be placed is based upon a computer-generated table with random numbers. For this, a categorical list in logical order will be created by an independent person before the start of the study. After being found eligible to start the study, the subject gets the following study number that is on the list. Basically, this entire randomization process is blinded and follows the concealed allocation procedures. During this process, it will safeguard that there are equal group sizes and an equal number of men and women in both groups (range 40/60% or 60/40% is accepted).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen hydrolysate (Experimental): 30 subjects will consume the protein hydrolysate daily for 4 weeks
  Interventions: Dietary Supplement: 10 g of collagen hydrolysate
- Placebo (Placebo Comparator): 30 subjects will consume the placebo daily for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 10 g of collagen hydrolysate — Before breakfast, participants consume 1 sachet every day for 4 weeks. The sachet contains 10-gram collagen protein hydrolysates + 5-gram erythritol and it has to be dissolved in 250 ml of water.
  Arms: Collagen hydrolysate
Dietary Supplement: Placebo — Before breakfast, participants consume 1 sachet every day for 4 weeks. The sachet contains 5-gram erythritol (placebo) and has to be dissolved in 250 ml of water.
  Arms: Placebo

SUMMARY:
The effects of a 10g/day collagen hydrolysate for a period of 4 weeks on glycemic control and cardiovascular health in a parallel design study using overweight/ obese men and women who are likely to have a disturbed lipid and glucose metabolism and increased risk to develop cardiovascular disease and/or Type- 2 diabetes.

DETAILED DESCRIPTION:
Food-derived bioactive peptides represent a source of health-enhancing components that have been reported to have cardiovascular health benefits in humans and may be incorporated in functional foods. Up till now studies using collagen hydrolysates particularly addressed issues around joint health, however, there are some preliminary indications that other health-related targets might be affected as well. We here propose to focus on the potential effects of collagen hydrolysates on glycemic control, and characteristics of the microcirculation, both important parameters for the assessment of future cardiovascular disease (CVD) risk.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40-75 years
* Men and women (in a ratio of 40/60 to 60/40)
* BMI between 25-35 kg/m2
* Serum total cholesterol < 8.0 mmol/L (further testing is recommended for excessive hyperlipidemia [serum total cholesterol ≥ 8.0 mmol/L] according to the Standard for cardiovascular risk management of the Dutch general practitioner's community [Nederlands Huisartsen Genootschap])
* Serum triacylglycerol < 4.5 mmol/L
* No current smoker
* No diabetic patients
* No familial hypercholesterolemia
* No abuse of drugs
* Not more than 4 alcoholic consumption per day with a maximum of 21 per week??
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* No use of medication known to treat blood pressure, lipid or glucose metabolism
* No use of an investigational product within another biomedical intervention trial within the previous 1-month
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, autoinflammatory diseases, and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or cardiovascular events, such as an acute myocardial infarction or cerebrovascular accident
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study, and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit
* Willing to comply to study protocol during the study
* Agree to take porcine / animal-derived supplements (i.e. collagen)
* Informed consent signed

Exclusion Criteria:

* Allergy or intolerance to collagen or collagen hydrolysates
* Serum total cholesterol ≥ 8.0 mmol/L
* Serum triacylglycerol ≥ 4.5 mmol/L
* Current smoker, or smoking cessation <12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 4 alcoholic consumptions per day or 21 per week
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use medication known to treat blood pressure, lipid, or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, autoinflammatory diseases, and rheumatoid arthritis
* Active cardiovascular diseases like congestive heart failure or cardiovascular events, such as an acute myocardial infarction or cerebrovascular accident
* Not willing to give up being a blood donor from 8 weeks before the start of the study, during the study, or for 4 weeks after completion of the study
* Not or difficult to venipuncture as evidenced during the screening visit
* Use of over-the-counter and prescribed medication or supplements, which may interfere with study measurements to be judged by the principal investigator;
* Use of oral antibiotics in 40 days or less prior to the start of the study;
* Blood donation in the past 3 months before the start of the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Chronic glucose metabolism | pre- intervention and during the fourth week of intervention.
  Measured by change in average daily glucose concentrations over a 15 hours period between waking up and going to bed 7:00-22:00 for three days, which is calculated based on the total area under the curve (tAUC) using a continuous glucose monitor.

SECONDARY OUTCOMES:
Lipid metabolism | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Measured by fasting serum, lipids and lipoproteins in all visits
Glucose metabolism | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Measured by fasting plasma glucose, and insulin in all visits
Low-grade inflammation | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Measured by inflammation plasma markers (Interleukin-6, Interleukin-8)
Postprandial glucose metabolism | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), and immediately after the intervention (visit 5)
  Following a high-fat, high-carb meal, measured by plasma glucose, insulin.
Postprandial triacylglyceride metabolism | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), and immediately after the intervention (visit 5)
  Following a high-fat, high-carb meal, measured by plasma triacylglyceride.
Quality of life questionnaire | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), during (at home), and immediately after the intervention (visit 5)
  Assessed with a 32-item questionnaire (including social, spiritual, emotional, cognitive, physical, activities of daily living, and integrated quality of life) Outcome Measures 1-5 (1= Bad, 2=Below Average, 3= Average, 4=Above Average, 5=Good .
Mood, degree of pleasantness and arousal | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), during (at home), and immediately after the intervention (visit 5)
  Assessed with the Affect grid
Perceived Stress Scale | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), during (at home), and immediately after the intervention (visit 5)
  Assessed using the Perceived Stress Scale Scale, a 10-item questionnaire that is used to determine individual stress levels experienced in the past weeks during daily activities. Scores ranging from 0-40 Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Cognitive performance | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), and immediately after the intervention (visit 5)
  Assessed with a validated neuropsychological test battery (Cambridge Neuropsychological Test Automated Battery) subjects will perform a neuropsychological test battery containing the anti-cue task (impulse control), the psychomotor vigilance test (sustained attention), the Attention Network Test, the N-Back task (working), the Rey Auditory Verbal Learning Task) (episodic memory), and the Trail Making Test (executive functioning).
Venular and arteriolar diameters | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), and immediately after the intervention (visit 5)
  Assessed via fundus photography
Office blood pressure | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Systolic and diastolic blood pressure measured by office blood pressure monitor in all visits
36-hours blood pressure profiles | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), and during the fourth week of intervention (visit 5)
  Systolic and diastolic blood pressure assessed via wearable blood pressure monitor
Sleep Quality | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), during (at home), and immediately after the intervention (visit 5)
  Assessed using the Pittsburgh Sleep Quality Index (PSQI) Consisting of 19 items. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by A total of seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Tumor necrosis factor alfa | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Measured by inflammation plasma markers Tumor necrosis factor alfa
C-reactive Protein | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Measured by inflammation plasma markers C-reactive Protein
Chronic glucose metabolism | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Measured by fasting plasma glycated hemoglobin A1c
Insulin sensitivity | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Measured by fasting calculated homeostasis model assessment of insulin resistance in all visits
C-peptide | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and during the fourth week of intervention (visit 4, and 5)
  Measured by fasting serum C-peptide
Cerebral blood flow (CBF) | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), and immediately after the intervention (visit 5)
  Measured using a DWL Multi-Dop T digital device (Compumedics Germany GmbH, Singen, Germany)

OTHER OUTCOMES:
Exploratory objective endothelial (dys)function markers | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and post intervention (visit 4, and 5)
  Measured by soluble endothelial molecule E-selectin, intercellular adhesion molecule-1, Circulating Vascular Cell Adhesion Molecule-1, and Monocyte Chemoattractant Protein-1 in al visits
Exploratory objective liver enzymes | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and post intervention (visit 4, and 5)
  Measured by liver enzymes (alanine aminotransferase, aspartate transaminase , gamma-glutamyltransferase , bilirubin)
Exploratory objective calculated insulin secretory function | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and post intervention (visit 4, and 5)
  Measured by The Homeostasis Model Assessment (HOMA) estimates steady state beta cell function (%B)
Exploratory objective plasma incretins / satiety hormones in fasting and postprandial conditions | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 3), and post intervention (visit 5)
  Following a high-fat, high-carb meal, measured by peptide YY , glucagon-like peptide-1, ghrelin.
Exploratory objective micro-albuminuria and kidney function | 2 weeks pre-intervention + 4 weeks intervention: Pre-intervention (visit 1,2 and 3), and post intervention (visit 4, and 5)
  Measured by estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, PhD, Principal Investigator — Chair of Nutrition and Movement Science Department
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manninen AH. Protein hydrolysates in sports and exercise: a brief review. J Sports Sci Med. 2004 Jun 1;3(2):60-3. eCollection 2004 Jun. PMID 24482579
- [Background] Thomson RL, Buckley JD. Protein hydrolysates and tissue repair. Nutr Res Rev. 2011 Dec;24(2):191-7. doi: 10.1017/S0954422411000084. Epub 2011 Nov 21. PMID 22098638
- [Background] Manninen AH. Protein hydrolysates in sports nutrition. Nutr Metab (Lond). 2009 Sep 28;6:38. doi: 10.1186/1743-7075-6-38. PMID 19785737
- [Background] de Campos Zani SC, Wu J, Chan CB. Egg and Soy-Derived Peptides and Hydrolysates: A Review of Their Physiological Actions against Diabetes and Obesity. Nutrients. 2018 Apr 28;10(5):549. doi: 10.3390/nu10050549. PMID 29710777
- [Background] Saleh L, Schrier NL, Bruins MJ, Steegers EAP, van den Meiracker AH, Visser W. Effect of oral protein hydrolysate on glucose control in patients with gestational diabetes. Clin Nutr. 2018 Jun;37(3):878-883. doi: 10.1016/j.clnu.2017.03.009. Epub 2017 Mar 16. PMID 28372849
- [Background] Power O, Nongonierma AB, Jakeman P, FitzGerald RJ. Food protein hydrolysates as a source of dipeptidyl peptidase IV inhibitory peptides for the management of type 2 diabetes. Proc Nutr Soc. 2014 Feb;73(1):34-46. doi: 10.1017/S0029665113003601. Epub 2013 Oct 17. PMID 24131508
- [Background] Benito-Ruiz P, Camacho-Zambrano MM, Carrillo-Arcentales JN, Mestanza-Peralta MA, Vallejo-Flores CA, Vargas-Lopez SV, Villacis-Tamayo RA, Zurita-Gavilanes LA. A randomized controlled trial on the efficacy and safety of a food ingredient, collagen hydrolysate, for improving joint comfort. Int J Food Sci Nutr. 2009;60 Suppl 2:99-113. doi: 10.1080/09637480802498820. Epub 2009 Feb 11. PMID 19212858
- [Derived] Chavez-Alfaro MA, Mensink RP, Joris PJ, Plat J. Effects of porcine-derived collagen hydrolysates on 24 h blood pressure profiles, markers for endothelial dysfunction and low-grade inflammation and the retinal vasculature in adults with overweight/obesity: a randomized, controlled trial. Food Funct. 2025 Dec 8;16(24):9562-9571. doi: 10.1039/d5fo01261a. PMID 41288414
- [Derived] Chavez-Alfaro MA, Mensink RP, Plat J. Effects of four-weeks porcine-collagen hydrolysate consumption on glucose concentrations, glycemic variability, and fasting/postprandial cardiometabolic risk markers in men and women with overweight or obesity: A randomized, controlled trial. Clin Nutr. 2025 Mar;46:60-71. doi: 10.1016/j.clnu.2025.01.018. Epub 2025 Jan 22. PMID 39889494